CLINICAL TRIAL: NCT03839615
Title: Assessment Of Poly Tetra Fluro Ethylene Membrane Versus Native Collagen Membrane With Guided Bone Regeneration In Atrophic Anterior Maxilla Using (1:1) Of Autogenous Bone And Xenograft Mixture (Randomized Clinical Trial)
Brief Title: Poly Tetra Fluro Ethylene vs Native Collagen Membrane for Gbr in Anterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, bassam ahmed abd elhameed alkholi, principle investigator (doctor), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GBR using ptfe vs collagen
Record Dates: First submitted 2018-12-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Missing Maxillary Anterior Teeth

STUDY DESIGN:
Who Masked: Investigator
Masking Description: each patient will be given a code by researcher and observer will be blind to which group this case belong
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided bone regeneration using ptfe (Active Comparator): Augmented anterior maxillary bone ridge using ptfe with 1:1 autogenous bone and xenograft mixture
  * Patients of both groups will be subjected to CBCT (diagnostic for upper arch).
  * Intra operative procedures (for both groups) followed by CBCT will be taken for every patient.
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  intervention:
  * Flap will be done.
  * In the group: bone decortication will be done using surgical round bur, autogenous bone will be harvested by trephine bur ,mixed 1:1 with anorganic bovine bone derived mineral mineral will be packed then covered at the defected area by a ptfe membrane which will be stabilized by tacks.
  Interventions: Procedure: guided bone regenerations
- collagen membrane (Experimental): * Local anesthesia will be given to the patient. intervention:
  * Flap will be done.
  * In the group: bone decortication will be done using surgical round bur, autogenous bone will be harvested by trephine bur ,mixed 1:1 with anorganic bovine bone derived mineral mineral will be packed then covered at the defected area by a native collagen membrane which will be stabilized by tacks.
  Interventions: Procedure: guided bone regenerations

INTERVENTIONS:
Procedure: guided bone regenerations — intra oral procedures.
  * Flap will be done.
  * In the study group: bone decortication will be done using surgical round bur, autogenous bone will be harvested by trephine bur ,mixed 1:1 with anorganic bovine bone derived mineral mineral will be packed then covered at the defected area by a native collagen membrane which will be stabilized by tacks.
  * In the control group: : bone decortication will be done using surgical round bur, autogenous bone will be harvested by trephine bur ,mixed 1:1 with anorganic bovine bone derived mineral and packed at the defected area then covered by a titanium reinforced polytetraflouroethelene membrane which will be stabilized by tacks.
  * The site will then be copiously irrigated with saline in preparation for closure.
  * The flap will then be closed using interrupted 4/0 resorbable sutures.

SUMMARY:
evaluation of amount of bone gained in the anterior maxilla using collagen membranes vs ptfe membrane while using a 1:1 mix of xenograft and autogenous bone

DETAILED DESCRIPTION:
The alveolar bone is formed during tooth eruption, and consists of maxillary and mandibular components that shape and support the alveolar sockets. When teeth are lost, alveolar atrophy occurs, ultimately resulting in a short and narrow alveolar ridge . Such changes in the alveolar bone have a significant effect on prosthetic restoration planning, and are particularly important for areas with esthetic requirements, such as the maxillary incisors. Since preservation of the alveolar bone after extraction makes implant placement and prosthetic restoration easier in the edentulous jaw, alveolar ridge preservation and reconstruction methods using various bone graft materials together with resorbable and non-resorbable membranes have been introduced in order to minimize the loss of alveolar bone after extraction.

Investigations of changes in the alveolar bone after extraction have frequently been performed through clinical measurements and radiographic analysis. In particular, after the extraction of a tooth with fracture or severe periodontitis, the alveolar bone shows severe horizontal and vertical atrophy. The reduction in the width of the alveolar ridge is more notable in the horizontal direction than in the vertical direction, and the buccal wall of the alveolar bone has been reported to undergo greater vertical atrophy than the lingual wall. Changes in the width of the alveolar ridge after extraction occur in a relatively short time, decreasing most rapidly within the first six months after extraction, followed by continual, slow bone resorption over the course of the rest of the patient's life .

When a tooth has been lost, the extent of alveolar bone resorption is affected by a range of factors, including the number of extracted teeth and bone walls, the bone density, the extent of alveolar bone loss, infection, and the presence or absence of adjacent teeth.

Dental implant has become a predictable treatment option, with excellent long-term results. However, the success of implant therapy depends on the amount of bone volume at the insertion site.Unfavorable local conditions may provide insufficient bone volume that negatively affects the prognosis of dental implants. Cawood and Howell in 1988 ranked the atrophy degree of edentulous jaws in six classes. Particularly, atrophies within class IV, also known as "knife-edge" ridges, present a serious horizontal defect, making challenging the placement of regular implants.

Many techniques have been developed to regenerate atrophic alveolar jaws for the placement of dental implants, performed either in combination with graft procedures or in second stage surgery after a period of healing. For many years, bone blocks represented the gold standard to reconstruct the alveolar ridge bone defects. This technique requires to harvest a wide amount of bone to rebuild the atrophic crest.(20). For this reason, bone blocks were often harvested from extra-oral sites with an higher morbidity. Moreover some problems can occur when a combined defects (horizontal and vertical) need to be treated. Guided bone regeneration (GBR) has been proposed as a possible alternative for patients with severe horizontal bone atrophy, to overcome the drawback of bone blocks techniques. To protect and prevent the invasion of the clot by nonosteogenic cells, maintaining an adequate biological space for the regeneration of bone tissue, the use of both non-resorbable or resorbable membranes, in combination with autologous or heterologous particulate bone have been proposed. Particulated autogenous bone can be mixed with bone substitutes to add more osteogenic factors.

Guided bone regeneration or GBR, and guided tissue regeneration or GTR are dental surgical procedures that use barrier membranes to direct the growth of new bone and gingival tissue at sites with insufficient volumes or dimensions of bone or gingiva for proper function, esthetics or prosthetic restoration.

GBR is similar to guided tissue regeneration (GTR) but is focused on development of hard tissues in addition to the soft tissues of the periodontal attachment. At present, guided bone regeneration is predominantly applied in the oral cavity to support new hard tissue growth on an alveolar ridge to allow stable placement of dental implants.

The first application of barrier membranes in the mouth occurred in 1982. in the context of regeneration of periodontal tissues via GTR, as an alternative to resective surgical procedures to reduce pocket depths.Barrier membrane is utilized in GBR technique to cover the bone defect and create a secluded space, which prevents the connective tissue from growing into the space and facilitates the growth priority of bone tissue.

Several surgical techniques via GBR have been proposed regarding the tri-dimensional bone reconstruction of the severely resorbed maxilla, using different types of bone substitutes that have regenerative, osseoinductive or osseoconductive properties which is then packed into the bony defect and covered by resorbable membranes. In cases where augmentation materials used are autografts or allografts the bone density is quite low and resorption of the grafted site in these cases can reach up to 30% of original volume. For higher predictability, nonresorbable titanium-reinforced d-polytetrafluoroethylene (d-PTFE) membranes-as a barrier against the migration of epithelial cells within the grafted site-are recommended.

Non-resorbable membranes retain their shape and structure in the tissues, requiring a second surgical procedure for removal, with consequent additional patient discomfort, and a raise in the costs and duration of the therapy. Non-resorbable membranes include: (i) expanded polytetrafluoroethylene (e-PTFE, Gore-Tex®); (ii) high-density polytetrafluoroethylene (d-PTFE) and (iii) titanium-reinforced expanded polytetrafluoroethylene (Ti-e-PTFE) membranes. The PTFE physico-chemical, thermal, and mechanical properties make it one of the most inert materials.The microstructure of e-PTFE consists of solid nodes interconnected by fine, highly oriented fibrils, providing a unique porous structure. The e-PTFE membranes, first used in 1984, have different structural features at both membrane sides.Effectiveness of e-PTFE membranes was investigated in numerous clinical studies, that confirmed their excellent biocompatibility, leading to a significant bone regeneration after 3- and 6-month healing period .However, drawbacks of e-PTFE membranes are (i) the need for a second surgical procedure and (ii) membrane stiffness that may result in soft tissue dehiscence (which is the cause of failure during the first 3 weeks after membrane implantation), allowing the exposure of the membrane to bacterial infection.

The d-PTFE membrane, developed in 1993, is a non-resorbable membrane, consisting of a high-density PTFE having submicron (0.2 μm) pores. The d-PTFE membranes do not require primary closure and preserve the full width of keratinized mucosa, producing an interesting advantage in respect to e-PTFE. Compared to e-PTFE membranes, the macroporosity of which enhances bacterial colonization upon exposure .the density of the d-PTFE membranes (i) prevents the infections as widely described by different authors .and (ii) makes membranes easy to be removed.

Titanium-reinforced barrier membranes were introduced (Cytoplast® TI-250 Titanium-Reinforced) by Jovanovic and Nevins . who reported the superior regenerative ability of these membranes in respect to the conventional e-PTFE ones. The titanium reinforcement provides mechanical support to the overlying soft tissue preventing its collapse into the defect. In addition, during the surgical procedure, titanium struts permit the surgeon to easily place the membrane under flaps with minimal dissection and flap reflection Native collagen membranes have rapid biodegradation by the enzymatic activity of macrophages and polymorphonuclear leucocytes occurs when using them. these membranes are well documented and have excellent results . they have good tissue integration and vascularization from periosteal side.there is a debate about what is more important biocompatibility or resorption time . The most important commercial collagen membrane is Bio-Gide®, which is based on Xenogenic collagen Type I form porcine skin and is characterized by a bilayered structure with a dense and a porous layer. The dense layer has a smooth surface able to avoid epithelial cell infiltration into bone defects, while the porous layer allows tissue integration.

ELIGIBILITY:
Inclusion Criteria:• Patients with atrophied anterior maxillary ridge area.

* Age: 18 years and older.
* Both sexes.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate bone augmentation.

Exclusion Criteria:

* • Heavy smokers more than 20 cigarettes per day.(32)

  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems.
  * Disorders to bone augmentation are related to history of radiation therapy to the head and neck neoplasia.
  * Pregnant or nursing women.
  * Patients with uncontrolled diabetes mellitus, rheumatoid arthritis or osteoporosis.
  * Patient with previous history of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — • human Patients with atrophied anterior maxillary ridge area.
Enrollment: 10 (Estimated)
Dates: Start 2019-02-26 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
amount of bone gained | 6 months
  using cbct 6 months after

SECONDARY OUTCOMES:
Bone area percentage | 6 months
  Histo-morphometric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univeristy, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tallgren A. The continuing reduction of the residual alveolar ridges in complete denture wearers: a mixed-longitudinal study covering 25 years. 1972. J Prosthet Dent. 2003 May;89(5):427-35. doi: 10.1016/s0022-3913(03)00158-6. No abstract available. PMID 12806317
- [Background] Pinho MN, Roriz VL, Novaes AB Jr, Taba M Jr, Grisi MF, de Souza SL, Palioto DB. Titanium membranes in prevention of alveolar collapse after tooth extraction. Implant Dent. 2006 Mar;15(1):53-61. doi: 10.1097/01.id.0000202596.18254.e1. PMID 16569962
- [Background] Kerr EN, Mealey BL, Noujeim ME, Lasho DJ, Nummikoski PV, Mellonig JT. The effect of ultrasound on bone dimensional changes following extraction: a pilot study. J Periodontol. 2008 Feb;79(2):283-90. doi: 10.1902/jop.2008.070289. PMID 18251642
- [Background] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Lekovic V, Camargo PM, Klokkevold PR, Weinlaender M, Kenney EB, Dimitrijevic B, Nedic M. Preservation of alveolar bone in extraction sockets using bioabsorbable membranes. J Periodontol. 1998 Sep;69(9):1044-9. doi: 10.1902/jop.1998.69.9.1044. PMID 9776033
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Camargo PM, Lekovic V, Weinlaender M, Klokkevold PR, Kenney EB, Dimitrijevic B, Nedic M, Jancovic S, Orsini M. Influence of bioactive glass on changes in alveolar process dimensions after exodontia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Nov;90(5):581-6. doi: 10.1067/moe.2000.110035. PMID 11077380
- [Background] Fiorellini JP, Howell TH, Cochran D, Malmquist J, Lilly LC, Spagnoli D, Toljanic J, Jones A, Nevins M. Randomized study evaluating recombinant human bone morphogenetic protein-2 for extraction socket augmentation. J Periodontol. 2005 Apr;76(4):605-13. doi: 10.1902/jop.2005.76.4.605. PMID 15857102
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Jahangiri L, Devlin H, Ting K, Nishimura I. Current perspectives in residual ridge remodeling and its clinical implications: a review. J Prosthet Dent. 1998 Aug;80(2):224-37. doi: 10.1016/s0022-3913(98)70116-7. PMID 9710828
- [Background] Pjetursson BE, Thoma D, Jung R, Zwahlen M, Zembic A. A systematic review of the survival and complication rates of implant-supported fixed dental prostheses (FDPs) after a mean observation period of at least 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:22-38. doi: 10.1111/j.1600-0501.2012.02546.x. PMID 23062125
- [Background] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791
- [Background] Esposito M, Grusovin MG, Coulthard P, Worthington HV. The efficacy of various bone augmentation procedures for dental implants: a Cochrane systematic review of randomized controlled clinical trials. Int J Oral Maxillofac Implants. 2006 Sep-Oct;21(5):696-710. PMID 17066630
- [Background] Simion M, Jovanovic SA, Tinti C, Benfenati SP. Long-term evaluation of osseointegrated implants inserted at the time or after vertical ridge augmentation. A retrospective study on 123 implants with 1-5 year follow-up. Clin Oral Implants Res. 2001 Feb;12(1):35-45. doi: 10.1034/j.1600-0501.2001.012001035.x. PMID 11168269
- [Background] Cawood JI, Howell RA. A classification of the edentulous jaws. Int J Oral Maxillofac Surg. 1988 Aug;17(4):232-6. doi: 10.1016/s0901-5027(88)80047-x. PMID 3139793
- [Background] Buser D, Ingimarsson S, Dula K, Lussi A, Hirt HP, Belser UC. Long-term stability of osseointegrated implants in augmented bone: a 5-year prospective study in partially edentulous patients. Int J Periodontics Restorative Dent. 2002 Apr;22(2):109-17. PMID 12019706
- [Background] Chiapasco M, Casentini P, Zaniboni M, Corsi E. Evaluation of peri-implant bone resorption around Straumann Bone Level implants placed in areas reconstructed with autogenous vertical onlay bone grafts. Clin Oral Implants Res. 2012 Sep;23(9):1012-21. doi: 10.1111/j.1600-0501.2011.02262.x. Epub 2011 Aug 9. PMID 22092480
- [Background] Urban IA, Jovanovic SA, Lozada JL. Vertical ridge augmentation using guided bone regeneration (GBR) in three clinical scenarios prior to implant placement: a retrospective study of 35 patients 12 to 72 months after loading. Int J Oral Maxillofac Implants. 2009 May-Jun;24(3):502-10. PMID 19587874
- [Background] Urban I, Caplanis N, Lozada JL. Simultaneous vertical guided bone regeneration and guided tissue regeneration in the posterior maxilla using recombinant human platelet-derived growth factor: a case report. J Oral Implantol. 2009;35(5):251-6. doi: 10.1563/AAID-JOI-D-09-00004.1. PMID 19882822
- [Background] Esposito M, Grusovin MG, Felice P, Karatzopoulos G, Worthington HV, Coulthard P. Interventions for replacing missing teeth: horizontal and vertical bone augmentation techniques for dental implant treatment. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD003607. doi: 10.1002/14651858.CD003607.pub4. PMID 19821311
- [Background] Wang HL, Boyapati L. "PASS" principles for predictable bone regeneration. Implant Dent. 2006 Mar;15(1):8-17. doi: 10.1097/01.id.0000204762.39826.0f. PMID 16569956
- [Background] Nyman S, Lindhe J, Karring T, Rylander H. New attachment following surgical treatment of human periodontal disease. J Clin Periodontol. 1982 Jul;9(4):290-6. doi: 10.1111/j.1600-051x.1982.tb02095.x. PMID 6964676
- [Background] Gottlow J, Nyman S, Karring T, Lindhe J. New attachment formation as the result of controlled tissue regeneration. J Clin Periodontol. 1984 Sep;11(8):494-503. doi: 10.1111/j.1600-051x.1984.tb00901.x. PMID 6384274
- [Background] Gottlow J, Nyman S, Lindhe J, Karring T, Wennstrom J. New attachment formation in the human periodontium by guided tissue regeneration. Case reports. J Clin Periodontol. 1986 Jul;13(6):604-16. doi: 10.1111/j.1600-051x.1986.tb00854.x. PMID 3462208
- [Background] 29.Horia Barbu, Monica Comăneanu, Mihai Bucur (Mar 2012).